CLINICAL TRIAL: NCT00587392
Title: Endoscopic Full-Thickness Plication for the Treatment of GERD: Long-Term Multicenter Results
Acronym: LTFU
Status: Completed | Type: Observational
Sponsor: NDO Surgical, Inc. (Industry)
Responsible Party: Bruce Gaumond, Associate Director, Clinical Affairs, NDO Surgical
Other Study IDs: 135-01928
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2007-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: Gastroesophageal Reflux Disease (GERD); Long-term follow-up (LTFU); Endoscopic Full-thickness Plication; Plicator
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Active NDO Endoscopic Full-thickness Plicator Procedure
  Interventions: Device: NDO Full-thickness Plicator

INTERVENTIONS:
Device: NDO Full-thickness Plicator — The NDO Full-thickness Plicator intervention was performed as part of the original open-label Plicator study as previously reported. This intervention did not take place as part of this long-term follow-up data collection study.

SUMMARY:
The purpose of this study was to gather long-term follow-up data on patients treated with the Plicator in a previous open-label multi-center study. Originally, 64 subjects were treated at seven U.S. sites. A subset of those patients were subsequently reassessed via symptom questionnaires in this long-term (60-month) follow-up analysis. The initial open-label study was completed and officially closed at the completion of 1-year follow-up. This current study was designed to collect long-term follow-up data on previously plicated subjects all of whom were recruited de novo from the original study population. Study endpoints were prospectively defined. The primary study objectives were to assess: reduction in GERD symptoms through analysis of the GERD Health Related Quality of Life (HRQL) questionnaire and the Gastrointestinal Symptom Rating Scale (GSRS); reduction in use of GERD medications, and change in overall physical and psychological health as measured by the Short Form Health Survey (SF-36).

ELIGIBILITY:
Inclusion Criteria (required prior to original treatment):

* History of heartburn or regurgitation for at least 6-months requiring maintenance daily anti-secretory therapy;
* esophageal manometry study demonstrating peristaltic amplitude >35mmHg and LES resting pressure >/=5mmHg;
* Increased esophageal acid exposure demonstrated through a 24-hour pH study.

Exclusion Criteria (required prior to original treatment):

* Erosive esophagitis (Savary-Miller grade III or IV);
* Barrett's esophagus;
* Esophageal stricture;
* Hiatal hernia >2cm;
* Persistent dysphagia, weight loss, esophageal bleeding, vomiting or gas-bloat
* Esophageal or gastric varices;
* Use of anticoagulants other than for cardiac prophylaxis
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously treated with the NDO Full-thickness Plicator in the original open-label study and who met the long-term Follow-up (LTFU) protocol inclusion and exclusion crieria were eligible for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction of GERD symptoms through analysis of GERD-Health Related Quality of Life (HRQL) questionnaire and Gastrointestinal Symptom Rating Scale (GSRS). | 3 and 5-years

SECONDARY OUTCOMES:
GERD Medication Use | 3 and 5-year
Improvement in overall health as measure by the short form Health Survey (SF-36). | 3 and 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Pleskow, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Boston MA; Simon Lo, MD, Principal Investigator — Cedars Sinai Medical Center, Lost Angeles, CA; Richard Rothstein, MD, Principal Investigator — Dartmouth Hitchcock Medical Center, Lebanon, NH; Christopher Gostout, MD, Principal Investigator — Mayo Clinic, Rochester, MN; Robert Hawes, MD, Principal Investigator — Medical University of South Carolina; Norman Marcon, MD, Principal Investigator — St. Michael's Hospital, Toronto, Ontario, Canada; Richard Kozarek, MD, Principal Investigator — Virginia Mason Medical Center, Seattle, WA
Locations (7):
- United States (6):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Medical University of South Carolina, Charleston, South Carolina
  - Virginia Mason Medical Center, Seattle, Washington
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Pleskow D, Rothstein R, Kozarek R, Haber G, Gostout C, Lembo A. Endoscopic full-thickness plication for the treatment of GERD: long-term multicenter results. Surg Endosc. 2007 Mar;21(3):439-44. doi: 10.1007/s00464-006-9121-8. Epub 2006 Dec 16. PMID 17180259
- [Result] Pleskow D, Rothstein R, Kozarek R, Haber G, Gostout C, Lo S, Hawes R, Lembo A. Endoscopic full-thickness plication for the treatment of GERD: Five-year long-term multicenter results. Surg Endosc. 2008 Feb;22(2):326-32. doi: 10.1007/s00464-007-9667-0. Epub 2007 Nov 20. PMID 18027032